CLINICAL TRIAL: NCT06901089
Title: Assessment of the Impact of Hip Manipulation on Muscle Strength and Stiffness as Well as Motor Functionality of Basketball Players During Training
Brief Title: Hip Manipulation in Basketball Players
Acronym: Manual Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: KB/96/2025
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-03

CONDITIONS: Manual Therapy; Manipulation; Muscles; Musculoskeletal System
MeSH Terms: interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Will be used: manipulation, placebo and exercise
  Interventions: Other: Manual therapy; Other: Placebo; Other: Exercise
- Group B (Placebo Comparator): Will be used: manipulation, placebo and exercise
  Interventions: Other: Manual therapy; Other: Placebo; Other: Exercise
- Group C (Active Comparator): Will be used: manipulation, placebo and exercise
  Interventions: Other: Manual therapy; Other: Placebo; Other: Exercise

INTERVENTIONS:
Other: Manual therapy — This technique involves a low-amplitude, high-velocity push on the hip joints with an additional two-second tension
Other: Placebo — This technique involves a low-amplitude, high-velocity push on the shoulder and elbow joints with an additional two-second tension
Other: Exercise — The following exercise will be performed: lunges

SUMMARY:
Currently, it is difficult to find studies in the literature assessing the impact of manual therapy on preventing lower limb injuries in basketball players, which may later translate into improved strength and balance in athletes, when planning training or therapy programming, e.g. in patients after ankle sprains.

ELIGIBILITY:
Inclusion Criteria:

* healthy persons aged 18,
* first league competitor,
* competitor who regularly competes in the league,
* expressing informed consent to participate in the study and undertakes to comply with track regulations and wear a helmet.

Exclusion Criteria:

* lack of volunteer consent,
* previous surgeries of the upper, lower limb and spine,
* other lower limb injuries in the last 6 months,
* pain limiting participation in the study,
* neurological diseases,
* connective tissue diseases.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of MVC. | The study will be conducted 3 times during one training session (before the intervention, after the intervention and after training). Each isometric muscle test lasts 3 seconds.
  Muscle EMG is an assessment of electrical characteristics during the test, the electrical source of which is the muscle membrane potential, and measured in μV.
Assessment of MVC. | The study will be conducted 4 times during one training session (before the intervention, after the intervention and after training).Each isometric muscle test lasts 3 seconds.
  Muscle EMG is an assessment of electrical characteristics during the test, which is measured by the repetition frequency of muscle motor unit discharges, which is measured in Hz, at the same time of the test.Time

SECONDARY OUTCOMES:
Assessment of proprioception. | The test will be performed three times during one training session (before the intervention, after the intervention, after the training). Each joint measurement will be performed at three settings: 15, 30, 45 degrees.
  Assessing proprioception is an assessment of the angular position of a joint and then an attempt to reproduce it, measured in degrees.
Y balance test | The test will be conducted three times during one training session (before the intervention, after the intervention, after training).
  Consists of the volunteer standing on one leg while simultaneously stretching the other lower limb in 3 different directions. These are: anterior, posteromedial and posterolateral.
Standing Long Jump Test | The test will be conducted 3 times during one training session (before the intervention, after the intervention, after the training). Each test is repeated 3 times.
  Attempt to jump as far as possible while landing on both feet without falling backwards. The distance will be measured and given in centimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- OSIR przy ul. Olimpijczyków Starogardzkich 1, Starogard Gdański, Poland

IPD SHARING:
Plan to Share IPD: No